CLINICAL TRIAL: NCT00213993
Title: Topical Antiperspirant for Prevention of Palmar-Plantar Erythrodysesthesia (Hand-Foot Syndrome) Associated With Capecitabine
Brief Title: Topical Antiperspirant for Hand-Foot Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2002-0487; CC-02308
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2007-12

CONDITIONS: Palmar-plantar Erythrodysesthesia
MeSH Terms: conditions — Hand-Foot Syndrome | interventions — Antiperspirants

ARMS (1):
- A (Experimental): antiperspirant topically to one foot once daily
  Interventions: Drug: antiperspirant

INTERVENTIONS:
Drug: antiperspirant — antiperspirant topically once daily to one foot

SUMMARY:
The objectives of this study are to evaluate the effectiveness of an antiperspirant in preventing or attenuating the severity of palmer-plantar erythrodysesthesia associated with the Food and Drug Administration (FDA)-approved doses of capecitabine. The hypothesis is that cytotoxic compounds in sweat will be prevented from being deposited in the skin and causing chronic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Has not previously received a regimen that includes 5-fluorouracil
* > 18 years old
* No known allergy or intolerance to Ban Unscented Roll-On Antiperspirant

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2006-10 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
reduction in palm and/or sole pain | after each of first four cycles of chemotherapy

SECONDARY OUTCOMES:
evaluation of utility of digital photography in the following palmar-plantar erythrodysesthesia (PPES) | after each of first four cycles of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Hutson, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States